CLINICAL TRIAL: NCT06271525
Title: Effect of Cupping Therapy on Nitric Oxide Level in Patients With Cervical Spondylosis
Acronym: CT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shady Abdelsattar Refaat (Other)
Responsible Party: Sponsor-Investigator, Shady Abdelsattar Refaat, principle investigator shady abdelsattar refaat, Cairo University
Organization: Cairo University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/002532
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Cervical Spondylosis
Keywords: cupping therapy; Cervical Spondylosis
MeSH Terms: conditions — Spondylosis | interventions — Cupping Therapy

STUDY DESIGN:
Intervention Model Description: cupping therapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cupping therapy (Experimental): patients with cervical spondylosis will receive cupping therapy one time per month for three months
  Interventions: Other: cupping therapy

INTERVENTIONS:
Other: cupping therapy — All the patients will be asked to be in a sitting position with both feet flat on the floor the cupping group will receive the cupping bloodletting at three acupuncture points (SI15, GB21, LI15) the medium size glass with a diameter of 4cm and a volume of 260ml. Each wet cupping treatment procedure will last about 20 min and will be conducted in five steps.
  1. -Primary sucking
  2. -Scarification 3- Bloodletting 4-Removal
  5 -Dressing

SUMMARY:
this study will be conducted to investigate the effect of cupping therapy on the nitric oxide level in patients with cervical spondylosis

DETAILED DESCRIPTION:
Cupping therapy is one of the oldest alternative medical procedures, along with acupuncture, with more than 3500 years of history to treat pain and various disorders. Cupping induces various biological responses that could be evoked by suction of the skin, About 5 to 10 minutes of cupping causes extravascular blood within the subcutaneous tissue and creates bruise-like marks. Therefore, cupping induces mild damage to a painful part of the body and accelerates healing by evoking the natural healing process. While this hypothesis is acceptable for some people, it might not be enough to change the minds of skeptics since cupping itself has no curative effects. Suppose the healing process after cupping can be accelerated by merging cupping with scientifically proven techniques. In that case, this new form of therapy might help to persuade skeptics of the efficacy of cupping. Integrative medicine, including acupuncture, dry needling, and cupping, is being used increasingly in the United States. evidence regarding their efficacy in the management of musculoskeletal conditions is heterogeneous and subject to several limitations. despite these limitations, acupuncture consistently is more effective than no treatment and is relatively safe. for chronic back pain, it is recommended as a first-line noninvasive therapy. for neck pain, acupuncture provides benefits when it is combined with other treatments. dry needling is similar to acupuncture and frequently is regarded as a form of acupuncture. sixty patients with cervical spondylosis will receive cupping therapy for three months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with (cervical spondylosis) from both sexes.
* Age range (24-60) in chronic stages.
* BMI from20-25 kg/m2.

Exclusion Criteria:

* Renal and hepatic patients.
* Anemia, hepatic disease, and dermatological diseases.
* Morbid obese patients if their BMI exceeds the 25 kg/m2 will be also excluded.
* the patients are taking any medications known to affect the pain level
* The patients have a systemic illness, dermatological problems, skin allergy, local ischemic problems

Ages: 24 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-20 (Estimated); Primary Completion 2024-05-20 (Estimated); Study Completion 2024-05-20 (Estimated)

PRIMARY OUTCOMES:
the nitric oxide level | up to three months
  Spectrophotometer device will be used to measure the level of nitric oxide

SECONDARY OUTCOMES:
cervical range of motion | up to three months
  electrogoniomter device will be used to assess cervical range of motion
pain intensity | up to three months
  visual analogue scale will be used to measure pain intensity. The VAS is a 100-mm horizontal line that may be used to quantify symptoms in a continuous fashion. It is easy to use and requires very little written language. Patients are instructed to indicate the intensity of their pain by marking on a line anchored by "no pain" on the left and "worst imaginable pain" on the right.